CLINICAL TRIAL: NCT03009032
Title: Immunological Effects of an Immunomodulatory Synbiotic Intervention at Advanced HIV Disease
Brief Title: Synbiotics in Advanced HIV Infection
Acronym: PROMALTIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Hospital San Carlos, Madrid (Other); Hospital Universitario 12 de Octubre (Other); Hospital Universitario La Paz (Other); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Hospital San Pedro de Logroño (Other); Hospital del Mar (Other)
Responsible Party: Principal Investigator, Sergio Serrano-Villar, MD, PhD, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14/016
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: HIV Infection Asymptomatic
Keywords: HIV; immunologic recovery; microbiota; prebiotics; probiotics; synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PMT25341 (Experimental): A mixture of prebiotics, probiotics, oligonutrients, essential aminoacids, omega-3 fatty acids
  Interventions: Dietary Supplement: PMT25341
- PLACEBO (Placebo Comparator): Lactose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PMT25341
  Arms: PMT25341
Dietary Supplement: Placebo — Lactose
  Arms: PLACEBO

SUMMARY:
Late diagnosed HIV-infected subjects show impaired immunological recovery resulting in a greater risk of clinical progression. Gut bacteria metabolism appears to impact immune recovery in HIV-infected subjects, and while nutritional interventions with prebiotics and probiotics seem to exert immunological effects, the clinical implications in this key population remain unknown. This is a pilot multicenter randomized placebo-controlled, double blind clinical trial in HIV-infected ART-naive subjects with <350 CD4 T cells/mm3 or AIDS. Participants will be randomized (1:1) to either the synbiotic nutritional supplement PMT25341 or placebo for 48 weeks, each in combination with first-line ART. Primary outcomes will be safety and immunological recovery. Secondary outcomes will include changes in fecal microbiota structure and plasma inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected ART-naive subjects with <350 CD4 T cells/mm3 or AIDS
* Initiating ART with any first-line regimen recommended in the Spanish GESIDA National Guidelines

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Type 1 or 2 diabetes
* End-stage renal disease
* Lactose intolerance
* Use of immunomodulatory drugs
* Neutrophil count <750cells/uL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From baseline through week 48
Changes in CD4+ T cell counts/uL | From baseline through week 48
Changes in CD8+ T cell counts/uL | From baseline through week 48
Changes in CD4/CD8 ratio | From baseline through week 48

SECONDARY OUTCOMES:
Microbiota composition: alpha-diversity | From baseline through week 48
Microbiota composition: Unifrac distances | From baseline through week 48
Microbiota composition: Canberra distances | From baseline through week 48
Changes in plasma soluble CD14 levels | From baseline through week 48
Changes in plasma hs-CRP levels | From baseline through week 48
Changes in plasma IFABP levels | From baseline through week 48
Changes in plasma lipoteichoic acid levels | From baseline through week 48
Changes in plasma kynurenine/tryptophan ratio | From baseline through week 48
Changes in percentage of HLADR+/CD38+ T cells | From baseline through week 48

IPD SHARING:
Plan to Share IPD: No